CLINICAL TRIAL: NCT06497218
Title: Smartphone-Based Neurobehavioral Assessments as a Diagnostic Aid in Autism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Blinklab Limited (Industry)
Collaborators: Mohammed VI National Center for the Disabled, Salé, Morocco (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13943
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: All subjects will undergo investigational diagnosis for ASD. Results will be compared to formal diagnosis by healthcare specialists.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children formally diagnosed with Autism Spectrum Disorder (Experimental): Children aged between 3 and 12 years with Autism Spectrum Disorder who received a formal DSM-5 diagnosis will be tested with Blinklab smart phone based diagnostic tool
  Interventions: Diagnostic Test: Blinklab diagnostic device

INTERVENTIONS:
Diagnostic Test: Blinklab diagnostic device — Blinklab is a non-invasive diagnostic device for Autism Spectrum Disorder

SUMMARY:
Retrospective case-control study to assess the diagnostic accuracy in autism spectrum disorder (ASD) of a new smartphone-based platform designed to conduct neurometric evaluations by measuring facial and behavioural reflexes.

DETAILED DESCRIPTION:
This is a retrospective multi-centre case-control study to measure sensorimotor anomalies linked to autism spectrum disorder (ASD) to assess the diagnostic accuracy of smartphone-based neurobehavioral evaluations. The primary objective of the study is to evaluate diagnostic accuracy of the smartphone-based assessments compared to a formal clinical diagnosis using machine learning algorithms.

Neurobehavioral testing will be performed using BlinkLab, a smartphone-based platform. The tests include general measurement of spontaneous and stimulus-evoked postural, head, facial, and vocal responses along with specific neurometric tests, including the acoustically evoked eyelid startle reflex (ASR), and tests that involve the modulation of the ASR, including prepulse inhibition (PPI) and habituation (HAB). Children required to participate in two consecutive 15-minute tests. During the experiment, the children will watch an audio-normalized movie while the trials containing the auditory stimuli will be delivered via headphones. For each trial, computer vision algorithms will be used to track and record the position of the participant's facial landmarks over time. The study will compare responses in children with ASD who received a formal DSM-5 based diagnosis prior to study inclusion and neurotypical children that had no formal psychiatric diagnoses.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals between the ages of 3 - 12 years old at the time of consent.
* Caregiver must be able to read, understand and sign the Informed Consent Form (ICF).
* Normal or corrected-to-normal vision with visual acuity sufficient to watch short videos.
* Hearing adequate to hear the auditory stimuli delivered via headphones.

Exclusion Criteria:

* Participants under 3 or over 12 years old.
* Severe hearing or visual impairment.
* Participants using medication that affects the nervous system (classified as ATC N0 medication, https://www.whocc.no).

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-10-16 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Device Sensitivity | at baseline
  Measure of the proportion of children truly having ASD who are correctly identified by the device as Positive for ASD relative to a formal DSM-5 diagnosis
Device Specificity | at baseline
  Measure of the proportion of children truly not having ASD (who had no prior psychiatric diagnosis) who are correctly identified by the device as Negative for ASD

SECONDARY OUTCOMES:
Screen Avoidance | at baseline
  The percentage of trials wherein the child was avoiding the smartphone's screen and camera
Anteroposterior Postural Stability | at baseline
  The child's anteroposterior postural stability
Head Rotations | at baseline
  The percentage of trials wherein the child was rotating their head
Headphone Touches | at baseline
  The percentage of trials wherein the child was touching the headphone
Mouth Opening | at baseline
  The size and timing of the child's mouth openings and closings
Vocalizations | at baseline
  The percentage of trials wherein the child was vocalizing and the corresponding time of occurrence
Acoustic Startle Response (ASR) | at baseline
  Difference in the amplitude of the eyelid ASR between the ASD and neurotypical children
Long-term habituation (long-term HAB) | at baseline
  Levels of habituation of the ASR over the course of the 15-minute test
Prepulse inhibition (PPI) | at baseline
  Reduction in the amplitude of the eyelid startle response due to prepulse stimuli
Short-term habituation (short-term HAB) | at baseline
  Habituation in the mean amplitude of eyelid startle responses over the course of the six startle pulses
Anticipatory eye blinks (AEB) | at baseline
  The anticipatory eye blinks (AEB) in predefined observation windows (OW) containing an omitted pulse. AEB were responses that were not triggered by the startle stimulus itself but rather by the expectation of an upcoming startle stimulus

CONTACTS AND LOCATIONS:
Locations (1):
- Mohammed VI National Center for the Disabled, Salé, Morocco

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boele HJ, Jung C, Sherry S, Roggeveen LEM, Dijkhuizen S, Ohman J, Abraham E, Uvarov A, Boele CP, Gultig K, Rasmussen A, Vinueza-Veloz MF, Medina JF, Koekkoek SKE, De Zeeuw CI, Wang SS. Accessible and reliable neurometric testing in humans using a smartphone platform. Sci Rep. 2023 Dec 18;13(1):22871. doi: 10.1038/s41598-023-49568-2. PMID 38129487